CLINICAL TRIAL: NCT01297387
Title: An Observational, Prospective Study Evaluating Feasibility of Peripheral Angioplasty in Diabetic Patients With Critical Limb Ischemia in C and D Obstructions of Transatlantic Inter-Society Consensus (TASC II).
Brief Title: Feasibility of Peripheral Angioplasty in Type D TASCII Lesions
Status: Completed | Type: Observational
Sponsor: IRCCS Multimedica (Other)
Responsible Party: Ezio faglia MD, Diabetic Foot Center IRCCS MultiMedica, Sesto San Giovanni Milano
Other Study IDs: 08/2007_Cardiovascolare
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes; Critical Limb Ischemia
Keywords: Diabetic Patients; Critical Limb Ischemia; Revascularization
MeSH Terms: conditions — Diabetes Mellitus; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Revascularization of limb ischemia: Procedure/Surgery
  Interventions: Other: PTA BPG procedure,

INTERVENTIONS:
Other: PTA BPG procedure, — Surgery PTA or BPG Procedure, according usual local clinical practice
  Other Names: Peripheral angioplasty

SUMMARY:
This observational prospective study will evaluate, according o usual local clinical practice, feasibility of endoluminal revascularization in diabetic patients with type C and D lesions, according to TASC II Criteria.

About 300 patients will be treated with usual revascularization procedure. Each patient will be followed at least 12 months to evaluate clinical outcome and limb salvage interventions.

DETAILED DESCRIPTION:
In 2000, the Trans Atlantic Inter-Society Consensus (TASC) stated that patients with CLI should be treated with revascularization, to provide sufficient blood flow to relieve the rest pain and heal skin lesions. TASC also suggested that the best procedure should avoid a general anaesthesia, pose a lesser systemic stress and have fewer serious complications.

All these considerations pose peripheral angioplasty (PTA) as the procedure of choice, when feasible.

Unfortunately, TASC Recommendations, published in 2000 and confirmed in 2007, use morphological criteria to define guidelines for the choice of revascularization procedure.

According to these recommendations, type C and D lesions, which comprise most serious stenosis and occlusions, affecting long tracts of vessels, are candidate to bypass interventions, more than PTA.

This choice was due to the first impression, then denied by BASIL study, that PTA could be affected by a reduced efficacy on limb salvage.

Diabetic Patients are characterized by high prevalence of long occlusions in crural arteries and this anatomical asset reduces, according to TASC II criteria, the feasibility of Bypass Graft (BPG) in a large number of such patients.

Our preliminary experience showed the feasibility of PTA in diabetic patients with Chronic Critical Limb Ischemia (CLI), with a high percentage of efficient revascularization, regardless of morphology and number of obstructions.

This study aims to evaluate outcomes after PTA procedure also in patients with lesions of 20 cm or longer in superficial femoral arteries or with "long lesions" in subpopliteal arteries.

All diabetic patients referring to our Diabetic Foot Centre either for foot lesions or rest pain will be assessed for the presence of Critical Limb Ischemia (CLI) according to TASC II Criteria.

These patients, according to usual local clinical practice, will undergo to angiographic evaluation and, if feasible, to peripheral angioplasty.

The peripheral pulses will be evaluated by palpation and auscultation with a continuous-wave Doppler technique, the ankle-pressure will be recorded, when assessable (foot arteries absent or not compressible because of medial calcifications), the transcutaneous oxygen tension (TcPO2) will be evaluated at the dorsum of the foot and a duplex scanning will be performed. In all patients with one reduced or absent foot pulse, TcPO2 < 50 mmHg, ankle-pressure < 70 mmHg, significant obstructions present at duplex scanning, an arteriography will be carried out. In all patient with obstruction > 50% of vessel diameter, PTA will be the first-choice revascularization procedure and will be performed in the same session of the angiographic study. In patients in whom PTA will not be feasible, a by-pass operation was considered. The patients in whom PTA or BPG were not possible, received a therapy with prostanoids or lumbar sympathectomy plus prostanoids, when possible. In patients in whom the therapies did not relieve the rest pain or the gangrene was extended above the Chopart joint, an above-the-ankle-amputation was proposed and performed.

PTA procedure PTA was considered indicated for angiographically documented obstructions greater than 50% of the vessel lumen. The procedures were performed under local anesthesia through antegrade puncture of the ipsilateral common femoral artery. If obstructions were present in the iliac trunk at duplex scanning, the puncture was performed by contralateral approach. Vessel recanalization was considered successful when direct flow was obtained in treated vessel, with no residual stenosis > 50% of vessel diameter along the artery.

BPG procedure The choice of proximal and distal BPG anastomoses depended on the angiographic picture and aimed at obtaining at least one patent foot artery. The inflow was optimized, when possible, by combining femoral-popliteal bypass and PTA of the iliac trunk. Moreover, also in view of a following distal angioplasty, the distal anastomosis was performed on the most suitable popliteal or tibial artery segment by using intraluminal clamping and microsurgical technique. The surgery has always been carried out under epidural anesthesia. The autogenous saphena vein was employed if present and in good condition. If venous conduit could not be used, alloplastic prosthetic material (polytetrafluoroethylene: PTFE) was employed and the peripheral below-the-knee anastomosis consisted of a venous cuff using the Miller's technique, or "composite" bypass with interposition of distal venous segments. The absence of an available saphena and an angiographic score of run off >7 on the Rutherford scale did not exclude any patient, who otherwise could be eligible only for a major amputation, from a revascularization with distal bypass.

Treatment of non revascularized patients Prostanoids (alprostadil-α-cyclodextrine 60-120 μgr/day) were infused intravenously on average 5 days before hospital discharge. When possible and accepted by the patients, lumbar sympathectomy was performed.

In all patients the pain change was recorded and the TcPO2 and ankle-pressure values were reassessed 5 days after the PTA, BPG, lumbar sympathectomy and medical therapy.

Limb salvage In patients complaining of rest pain without foot ulcer, the disappearance of pain was considered to be a successful limb salvage. In patients with foot ulcer we considered limb salvage successful when the ulcer was healed and plantar stand was maintained, even when achieved by tarsal-metatarsal amputation and the patient is able to walk without crutches or artificial leg. Conversely, any above-the-ankle amputation was considered a failure. Limb salvage was considered early when pain disappeared and ulcer healed in 30 days after hospital admission.

Follow-up After hospital discharge All the patients with foot ulcer were examined weekly until ulcer healing. All patients were provided with extra-deep rocker shoes with soft thermoformable leather and customized insoles.

Evidence of PTA restenosis was assessed clinically only, based on pain reappearance or ulcer recurrence. In these situations ankle-pressure and TcPO2 were reassessed and duplex scanning was performed (22). If ankle pressure and TcPO2 were significantly worse (<15% of the post-PTA value) and Duplex scanning was positive, the patient underwent a repeated angiographic evaluation and a further PTA, if possible. Morphological restenosis was not investigated: in absence of rest pain or ulcer reappearance we do not perform any revascularization (23), therefore we consider the morphological restenosis clinically irrelevant.

BPG treated patients were followed with vascular surgery protocol (24). The graft patency was assessed with clinical examination and ultrasound study at 30 days, 3,6,12 months and thereafter every 6 months. Pulse systolic velocity and anastomosis morphology were assessed by ultrasound study. Finally, inflow is compared with pre-operative condition.

For every invasive treatment (PTA, BPG, sympathectomy, surgical operation on the foot) the written informed consent form was proposed and obtained from the patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult diabetic patients type 1 or 2
* Chronic critical ischemia as defined by TASC 2007 criteria (pain at rest, and/or ulcer or gangrene due to arteriopathy: transcutaneous oximetry < 30 mmHg or pressure on the ankle < 70 mmHg)

Exclusion Criteria:

* Cancer with adverse prognosis in months, or chemotherapeutic treatment
* Ongoing or planned pregnancy
* Lack of consent to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with critical limb ischemia
Sampling Method: Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2009-01; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ezio Faglia, MD, Principal Investigator — Diabetic Foot Centre IRCCS MultiMedica
Locations (1):
- Diabetic Foot Center IRCCS MultiMedica, Sesto San Giovanni, Milano, Italy